CLINICAL TRIAL: NCT06204952
Title: Effectiveness of Joins® for Managing Lumbar Facetogenic Pain: A Prospective, Randomized, Double-blind, Placebo-controlled, Pilot Study
Brief Title: Effectiveness of Joins® for Managing Lumbar Facetogenic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeeyoun Moon (Other)
Responsible Party: Sponsor-Investigator, Jeeyoun Moon, Professor, Seoul National University
Organization: Seoul National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2309-118-1470
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Facet Joint Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Take placebo drug 1T tid for 12 weeks.
  Interventions: Drug: Placebo
- Test drug (Active Comparator): Take Joins®(Clematidis Radix,Trichosanthes Root,Prunella Spike Extract) 1T tid for 12 weeks.
  Interventions: Drug: Joins®(Clematidis Radix,Trichosanthes Root,Prunella Spike Extract)

INTERVENTIONS:
Drug: Joins®(Clematidis Radix,Trichosanthes Root,Prunella Spike Extract) — In patients with facet joint syndrome, Joins® (Clematidis Radix, Trichosanthes Root, Prunella Spike Extract) is administered at a dosage of 1 tablet three times a day for 12 weeks.
  Arms: Test drug
Drug: Placebo — In patients with facet joint syndrome, placebo drug is administered at a dosage of 1 tablet three times a day for 12 weeks.
  Arms: Placebo

SUMMARY:
Obtain informed consent from patients with lumbar facet joint syndrome and, after enrollment, randomly assign them to Group A (Joins®) or Group B (Placebo). According to the allocation in each group, participants are instructed to take Joins® 200mg 1 tablet three times a day or placebo 1 tablet three times a day from day 1. Research subjects visit at 4-week intervals a total of 3 times (4 weeks, 8 weeks, 12 weeks) to collect various measurement variables. Both the test and control groups are observed during the period of taking the investigational medication without any changes or additional facet joint-related procedures (medial branch block, facet joint block). Acetaminophen is allowed as a rescue medication.

DETAILED DESCRIPTION:
First Visit (-4 weeks to 0 weeks, Screening Visit)

Check the most severe and average 11-point NRS pain scores in the last 24 hours, as well as the current 11-point NRS pain score. (To be eligible for the study, the average 11-point NRS pain score in the last 24 hours should be 4 or higher.) Conduct demographic survey, confirm concurrent medications and treatments, review medical and surgical history, and perform a physical examination. Measure vital signs. Conduct laboratory tests, and for fertile women, perform a pregnancy test. Perform lumbar X-ray examination. Perform lumbar MRI examination. (This examination can be arranged in advance at an external hospital for the purpose of this study.)

Second Visit (0 weeks, Enrollment and Randomization Visit)

After confirming the laboratory tests and lumbar X-ray conducted during the last visit, proceed with randomization only if deemed eligible for the study. Measure vital signs. Check the most severe and average 11-point NRS pain scores in the last 24 hours, as well as the current 11-point NRS pain score. Self-assess the questionnaires collected during this visit. Oswestry Disability Index (ODI), PainDETECT, GAD-7, EQ-5D Prescribe the test drug and placebo. Subjects will administer the test drug as follows from the day after the visit:

Placebo Group: Administer placebo orally three times a day, one tablet per dose, for 12 weeks.

Test Group: Administer Joins® 200 mg orally three times a day, one tablet per dose, for 12 weeks.

Confirm concurrent medications and treatments, and check for adverse reactions.

Third and Fourth Visits (4 weeks/8 weeks, Treatment Visits)

Measure vital signs. Check the most severe and average 11-point NRS pain scores in the last 24 hours, as well as the current 11-point NRS pain score. Self-assess the questionnaires collected during this visit. Oswestry Disability Index (ODI) Subjects return the remaining medication after administration. Confirm compliance and prescribe new test drugs. Confirm concurrent medications and treatments, and check for adverse reactions.

Fifth Visit (12 weeks, End of Treatment Visit)

Measure vital signs. Check the most severe and average 11-point NRS pain scores in the last 24 hours, as well as the current 11-point NRS pain score. Self-assess the questionnaires collected during this visit. Oswestry Disability Index (ODI), PainDETECT, GAD-7, EQ-5D, PGIC, Satisfaction with Investigational Medication Subjects return the remaining medication after administration.

Confirm compliance. Confirm concurrent medications and treatments, and check for adverse reactions. Conduct laboratory tests, and for fertile women, perform a pregnancy test.

Sixth Visit (13 weeks, Post-Treatment Follow-up Visit)

Measure vital signs. Check for adverse reactions. Conduct laboratory tests, and for fertile women, perform a pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 19 and 80 years of age
2. Those diagnosed with lumbar facet joint syndrome through diagnostic posterior medial limb block
3. Those with an average 11-point numeric rating scale (NRS) of 4 or more for back pain over the past 24 hours
4. Those who voluntarily decided to participate in the study and gave written consent

Exclusion Criteria:

1. Patient refusal
2. If the main cause of the current back pain is infectious spondyloarthrosis/arthropathy, ankylosing spondylitis, or stenosis, or if the patient complains or shows signs of local neurological symptoms (e.g., decreased motor power in the lower extremities) due to the underlying disease.
3. Patients with moderate to severe lumbar instability requiring surgery
4. Cognitive decline to the point where the numeric pain rating (NRS) cannot be understood.
5. Severe cardiovascular disease (Systolic BP >=160 mm Hg or diastolic BP >=100 mm) or liver (AST/APT increased more than twice normal) or kidney disease (GFR<60 mL/min/1.73 m2) A person with teeth
6. Those with systemic infection or spinal infection
7. Those who are allergic to clinical trial drugs or their ingredients
8. People with genetic problems such as galactose intolerance, lactase deficiency, or glucose-galactose malabsorption
9. If you are pregnant or breastfeeding. For women of childbearing potential, those who are unwilling to use a reliable method of contraception during the administration period and for more than 4 weeks after the last administration of the investigational drug

   * Women who have had menarche and have not reached postmenopausal status (≥12 months of consecutive amenorrhea without an identified cause other than menopause) and who have not undergone surgical sterilization (ovarian and/or hysterectomy) are considered women of childbearing potential.
   * You must remain abstinent (abstain from sexual intercourse with the opposite sex) or use two medically acceptable forms of contraception. One method of contraception with a low failure rate, defined as less than 1% per year (e.g., oral contraceptives or intrauterine device), and a medically acceptable second method, such as spermicide and condom use by the male partner, should be used. Barrier methods alone are not permitted. Male subjects should use condoms and spermicides during sexual intercourse, and female contraceptive partners should also be careful to use at least one additional method of contraception with a low failure rate as defined above.
   * The reliability of sexual abstinence must be evaluated considering the clinical trial period and the test subject's preferred daily lifestyle habits. Periodic abstinence (e.g., date, ovulation, symptom-temperature, or post-ovulation abstinence) and external ejaculation are not acceptable methods of contraception.
10. Those with malignant tumor in the lumbar region
11. Those who have previously undergone lumbar surgery or are scheduled to undergo spine surgery within 12 weeks after screening
12. Subjects who participated in other clinical trials within 6 months before the first administration of the investigational drug
13. Other people who are not suitable for this clinical trial according to the researcher's judgment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-06-22 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Comparison between two groups of change (%) in 11-point NRS | 12 weeks after the baseline
  Comparison between two groups of change (%) in 11-point NRS at 12 week visits compared to baseline

SECONDARY OUTCOMES:
Comparison between two groups of change (%) in 11-point NRS | 4 weeks and 8 weeks after the baseline
  Comparison between two groups of change (%) in 11-point NRS at 4- and 8-week visits compared to baseline
Within-group comparison of change (%) in 11-point NRS | 4 weeks, 8 weeks and 12 weeks after the baseline
  Within-group comparison of change (%) in 11-point NRS at 4-, 8-, and 12-week visits compared to baseline
Oswestry disability index (ODI) | 4 weeks, 8 weeks and 12 weeks after the baseline
  Oswestry disability index (ODI): Comparison of changes (%) and absolute values at 4-, 8-, and 12-week visits compared to baseline between and within groups (0-45)
PainDETECT/GAD-7/EQ-5D | 4 weeks, 8 weeks, and 12 weeks after the baseline
  PainDETECT/GAD-7/EQ-5D: Comparison of changes (%) and absolute values at the 12-week visit compared to baseline between groups and by time point within groups (0-45)
Patient's Satisfaction of pain | 12 weeks after the baseline
  Satisfaction with PGIC and clinical investigational drugs (%)
Patient's medication | 12 weeks after the baseline
  Patient's medication (comparison between groups regarding stable regimen, number of rescue medications taken, and dose taken)

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manchikanti L, Pampati V, Fellows B, Bakhit CE. Prevalence of lumbar facet joint pain in chronic low back pain. Pain Physician. 1999 Oct;2(3):59-64. PMID 16906217
- [Background] Manchikanti L, Boswell MV, Singh V, Pampati V, Damron KS, Beyer CD. Prevalence of facet joint pain in chronic spinal pain of cervical, thoracic, and lumbar regions. BMC Musculoskelet Disord. 2004 May 28;5:15. doi: 10.1186/1471-2474-5-15. PMID 15169547
- [Background] Cohen SP, Raja SN. Pathogenesis, diagnosis, and treatment of lumbar zygapophysial (facet) joint pain. Anesthesiology. 2007 Mar;106(3):591-614. doi: 10.1097/00000542-200703000-00024. PMID 17325518
- [Background] Enthoven WT, Roelofs PD, Deyo RA, van Tulder MW, Koes BW. Non-steroidal anti-inflammatory drugs for chronic low back pain. Cochrane Database Syst Rev. 2016 Feb 10;2(2):CD012087. doi: 10.1002/14651858.CD012087. PMID 26863524
- [Background] Abraham NS, Castillo DL, Hartman C. National mortality following upper gastrointestinal or cardiovascular events in older veterans with recent nonsteroidal anti-inflammatory drug use. Aliment Pharmacol Ther. 2008 Jul;28(1):97-106. doi: 10.1111/j.1365-2036.2008.03706.x. Epub 2008 Apr 7. PMID 18397385
- [Background] Lung YB, Seong SC, Lee MC, Shin YU, Kim DH, Kim JM, Jung YK, Ahn JH, Seo JG, Park YS, Lee CS, Roh KJ, Han CK, Cho YB, Chang DY, Kwak WJ, Jung KO, Park BJ. A four-week, randomized, double-blind trial of the efficacy and safety of SKI306X: a herbal anti-arthritic agent versus diclofenac in osteoarthritis of the knee. Am J Chin Med. 2004;32(2):291-301. doi: 10.1142/S0192415X04001941. PMID 15315266
- [Background] Choi JH, Choi JH, Kim DY, Yoon JH, Youn HY, Yi JB, Rhee HI, Ryu KH, Jung K, Han CK, Kwak WJ, Cho YB. Effects of SKI 306X, a new herbal agent, on proteoglycan degradation in cartilage explant culture and collagenase-induced rabbit osteoarthritis model. Osteoarthritis Cartilage. 2002 Jun;10(6):471-8. doi: 10.1053/joca.2002.0526. PMID 12056850
- [Background] Kim JI, Choi JY, Kim KG, Lee MC. Efficacy of JOINS on Cartilage Protection in Knee Osteoarthritis: Prospective Randomized Controlled Trial. Knee Surg Relat Res. 2017 Sep 1;29(3):217-224. doi: 10.5792/ksrr.17.004. PMID 28854768
- [Background] Sae-Jung S, Jirarattanaphochai K. Outcomes of lumbar facet syndrome treated with oral diclofenac or methylprednisolone facet injection: a randomized trial. Int Orthop. 2016 Jun;40(6):1091-8. doi: 10.1007/s00264-016-3154-y. Epub 2016 Mar 18. PMID 26987980
- [Background] Cohen SP, Moon JY, Brummett CM, White RL, Larkin TM. Medial Branch Blocks or Intra-Articular Injections as a Prognostic Tool Before Lumbar Facet Radiofrequency Denervation: A Multicenter, Case-Control Study. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):376-83. doi: 10.1097/AAP.0000000000000229. PMID 26066382